CLINICAL TRIAL: NCT01641276
Title: Identification of Specific Modulation Frequencies in Hepatitis B Carriers With and Without Hepatocellular Carcinoma
Acronym: THBC-HSL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Frederico Perego Costa, Attending physician, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 02621512.3.0000.5461
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis; Hepatocellular Carcinomas
Keywords: biofeedback response
MeSH Terms: conditions — Hepatitis; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hepatitis (Experimental): hepatitis B carriers patients
  Interventions: Device: Low intensity amplitude-moduled electromagnetic fields
- hepatocellular carcinoma patients (Experimental): hepatites B carriers patients with associated hepatocellular carcinoma
  Interventions: Device: Low intensity amplitude-moduled electromagnetic fields

INTERVENTIONS:
Device: Low intensity amplitude-moduled electromagnetic fields — Patients in each arm will be exposed to 30 min of amplitude-moduled low intensity electromagnetic fields only one time.
  Other Names: TheraBionic; OncoBionic P1

SUMMARY:
The propose of this study is to identification of a group of specific amplitude-modulated frequencies of low intensity electromagnetic fields that is associated with biofeedback upon exposure to in patients with hepatitis B carries with or without hepatocellular carcinoma.

DETAILED DESCRIPTION:
Patients will be exposed by different specific amplitude-modulated frequencies of low intensity electromagnetic fields for 30 min. During the exposure, autonomic response with be recorded in order to identify biofeedback response. Differences in group of frequencies is expected in patients with hepatitis B carries with or without hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* hepatitis B carriers patients
* hepatitis B carriers patients with hepatocellular cancer patients

Exclusion Criteria:

* other tumor types
* other hepatitis types

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Identification of different group of specific frequencies of modulation in hepatitis B carriers with and without hepatocellular carcinoma associated with biofeedback response | within 10 min of exposure
  biofeedback response will be monitored

SECONDARY OUTCOMES:
Characterization of differences biofeedback response in hepatitis B carriers with and without hepatocellular carcinoma | within 10 minutes of exposure
  Representation of autonomous response during the exposure of specific frequencies of modulation

CONTACTS AND LOCATIONS:
Overall Officials: Frederico P Costa, MD, Principal Investigator — Hospital Sirio-Libanes
Locations (1):
- Hospital Sírio Libanês, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Results of a phase II study on patients with hepatocellular carcinoma — http://www.nature.com/bjc/journal/v105/n5/full/bjc2011292a.html